CLINICAL TRIAL: NCT04079270
Title: A Phase 2 Single-blinded Randomized Study of Algorithm-based Personalized Nutrition Intervention Compared to Standard Diet Intervention in Patients Treated With Endocrine Therapy for Early Stage, Hormone Receptor Positive Breast Cancer
Brief Title: The Breast Cancer Personalized Nutrition Study
Acronym: BREACPNT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Principal Investigator, Dr. Einav NiliGal-Yam, Deputy Head, Breast Cancer Institute, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SMC- 5725-18
Record Dates: First submitted 2019-07-07; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer
Keywords: Weight gain; Endocrine treatment
MeSH Terms: conditions — Breast Neoplasms; Weight Gain | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized algorithm-based diet (Experimental): The intervention arm will be an 'algorithm-based' arm in which patients will receive personally tailored dietary recommendations, based on their microbiome, and other clinical data such as blood tests and lifestyle features.
  Interventions: Other: Nutrition intervention
- standard Mediterranean low-fat diet (Active Comparator): The control arm will receive nutritional recommendations according to the standard Israeli dietary approach Mediterranean-style low-fat diet.
  Interventions: Other: Nutrition intervention

INTERVENTIONS:
Other: Nutrition intervention — The diet recommendations will be provided by a certified dietitian. Participants will be asked to document their food intake and daily activities including exercise and sleep using a dedicated smartphone app throughout the intervention period.

SUMMARY:
The Breast Cancer Personalized Nutrition (BREACPNT) study will evaluate the effect of a microbiome based personalized diet intervention on control of weight gain, glycemic response, disease outcome and various biomarkers in hormone receptor early breast cancer patients receiving adjuvant endocrine treatment.

DETAILED DESCRIPTION:
Weight gain is a common incident in breast cancer survivors. As many as 50-96% of women experience weight gain during treatment. Endocrine treatment was identified as a risk factor for weight gain in several studies. Hence, weight management for breast cancer survivors is important for increasing adherence to therapy and lowering recurrence risk.

The essential role of the gut microbiota in modulating immune and metabolic functions in health and disease is increasingly recognized. Particularly in breast cancer (BC), diet plays an important role in creating a microbiome environment involved in estrogens metabolism. The microbiome directly affects the body's response to food.

The Personalized Nutrition Project, conducted in the Weizmann Institute of Science, showed that individuals vary greatly in their glycemic response to the same food, influenced by the involvement of functional microbial pathways. This study yielded an algorithm capable of accurately predicting personalized postprandial glycemic response (PPGR) to arbitrary meals. These results suggest that individually tailored dietary interventions help maintain normal blood glucose levels and influence microbiome diversity, which, in turn, can control weight changes.

In this phase 2 randomized trial, 200 Hormone receptor (HR) positive breast cancer patients, eligible for adjuvant endocrine therapy will be recruited to the study. Upon recruitment, subjects will provide a stool sample for microbiome analysis and will undergo continuous glucose monitoring for 2 weeks. Thereafter, patients will be randomly assigned in a 1:1 ratio to receive a personalized diet recommendation or a standard low-fat diet for 6 months. The algorithm is based on patients' microbiome analyses and other blood tests. Patient clinical records will be followed 2-3 times yearly for 5 years for DFS and BC recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with stage 1-3 breast cancer, who underwent surgery, have finished their neo/adjuvant chemotherapy and radiotherapy if these were indicated and are treated with adjuvant endocrine therapy (either Tamoxifen or Aromatase inhibitor +/- GNRH agonists).
* Patients are at least 60 days after finishing their last non-endocrine oncology treatment (i.e. definitive surgery, radiation or chemotherapy - whichever is last), have received at least 30 days of endocrine therapy ( tamoxifen or aromatase inhibitor) but no more than 24 months.
* Patients treated with neoadjuvant endocrine therapy are eligible provided they had undergone surgery, are least 60 days post their last non endocrine therapy (definitive surgery or radiation and chemotherapy, if these were indicated), are continuing their endocrine therapy but did not receive more than 24 months post-surgery.
* Are willing to work with smart phone application

Exclusion Criteria:

* Oral Antibiotics/antifungal use in the previous 3 months to profiling stage ( these patients will be able to join the study at a later point)
* Use of anti-diabetic and/or weight-loss medication
* BMI<18.5
* People under another diet regime and/or a dietitian consultation/another study?
* Pregnancy, breast feeding
* HIV carriers, Cushing syndrome, Chronic Kidney Disease, acromegaly, hyperthyroidism, liver cirrhosis
* Psychiatric disorders (Schizophrenia, Bipolar Disorder)
* Known diagnosis of IBD (inflammatory bowel diseases)
* Patients that underwent Bariatric surgery
* Known Alcohol or substance abuse
* Known Diagnosis of diabetes

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-07-17 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of a personalized diet compared to a standard low fat diet to control body mass as measured by changes in body mass. | 6 months intervention period.
  Body weight changes will be defined as the net body weight gained/lost

SECONDARY OUTCOMES:
To evaluate the efficacy of the personalized diet compared to a standard low fat diet to control glycemic response. | 6 months intervention period.
  glycemic response control measured by the area under the glucose curve (AUC) during continuous glucose monitoring (CGM) period.

OTHER OUTCOMES:
Evaluate disease outcome as measured by disease free survival in study subjects. | 5 years
  Disease free survival (DFS), years
To investigate microbiome composition and modulation during the diet intervention period and assess if there are differences in modulations between the personalized diets as compared to the standard diet | 6 months intervention period.
  changes in microbiome compositions

CONTACTS AND LOCATIONS:
Overall Officials: Gal-Yam, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request .
Supporting Information: Study Protocol, SAP
Time Frame: 12 months after publication
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents

REFERENCES:
- [Background] Zeevi D, Korem T, Zmora N, Israeli D, Rothschild D, Weinberger A, Ben-Yacov O, Lador D, Avnit-Sagi T, Lotan-Pompan M, Suez J, Mahdi JA, Matot E, Malka G, Kosower N, Rein M, Zilberman-Schapira G, Dohnalova L, Pevsner-Fischer M, Bikovsky R, Halpern Z, Elinav E, Segal E. Personalized Nutrition by Prediction of Glycemic Responses. Cell. 2015 Nov 19;163(5):1079-1094. doi: 10.1016/j.cell.2015.11.001. PMID 26590418
- [Background] Nyrop KA, Williams GR, Muss HB, Shachar SS. Weight gain during adjuvant endocrine treatment for early-stage breast cancer: What is the evidence? Breast Cancer Res Treat. 2016 Jul;158(2):203-17. doi: 10.1007/s10549-016-3874-0. Epub 2016 Jun 24. PMID 27342454
- [Derived] Rein MS, Dadiani M, Godneva A, Bakalenik-Gavry M, Morzaev-Sulzbach D, Vachnish Y, Kolobkov D, Lotan-Pompan M, Weinberger A, Segal E, Gal-Yam EN. BREAst Cancer Personalised NuTrition (BREACPNT): dietary intervention in breast cancer survivors treated with endocrine therapy - a protocol for a randomised clinical trial. BMJ Open. 2022 Nov 21;12(11):e062498. doi: 10.1136/bmjopen-2022-062498. PMID 36410828